CLINICAL TRIAL: NCT01308099
Title: Assessment of Vascular Endothelial Function in Postural Tachycardia Syndrome (POTS)
Brief Title: Assessment of Vascular Endothelial Function in Postural Tachycardia Syndrome
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Alfredo Gamboa, Research Assistant Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 091332
Record Dates: First submitted 2011-02-18; First posted 2011-03-03 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Postural Tachycardia Syndrome
Keywords: POTS; Vascular Endothelial Function
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Blood Pressure

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POTS & Controls: Participants will have a physical prior to the study day and collect urine for 24 hours.
  On the study day the following procedures take place:
  After blood samples taken (about 2 tbsp), the subject will lie down. A blood pressure cuff will be placed on one arm and small probes on one finger on both hands. The arm blood pressure cuff will be inflated 60 points above the highest number on your normal blood pressure for five minutes. The blood pressure and forearm blood flow will be recorded. At the end of 5 minutes, the cuff will be released and the measurements of blood pressure and calf blood flow will be repeated. The brachial artery diameter and flow will be measured at baseline, during cuff inflation and for 3 minutes after deflation.
  The study lasts about 2 hours.
  Interventions: Device: Blood Pressure and Blood Flow

INTERVENTIONS:
Device: Blood Pressure and Blood Flow — A blood pressure cuff will be placed on one arm and small probes on one finger on both hands. The probes also measure blood pressure. After 10 minutes, the arm blood pressure cuff will be inflated. The cuff will stay inflated for 5 minutes, then the air will be let out. A cuff will be place above the left calf and the left knee. The subject will lie quietly for 9 minutes, then blood pressure and calf blood flow will be measured for one minute. the lower leg cuff will be inflated after 1 minute, then the cuff will be deflated. The blood pressure and forearm blood flow will be recorded. Next, the cuff on the upper leg will be inflated for 5 minutes then, it will be released and the measurements of blood pressure and calf blood flow will be repeated.
  The study lasts about 2 hours.
  Other Names: Pulsitile Arterial Tonometry Protocol (PAT)

SUMMARY:
The purpose of this study is to see if people with Postural Tachycardia Syndrome (POTS) have different levels of certain chemicals in their blood than people who don't have POTS. This study will test whether the blood vessels of people with POTS will react differently to certain tests than people without POTS.

The hypothesis of the study is:

Patients with POTS will have vascular endothelial dysfunction compared with control subjects.

ELIGIBILITY:
Inclusion Criteria:

ALL:

* Ages between 18-60 years old
* Male and female subjects are eligible
* Able and willing to give informed consent

Additional criteria for POTS:

* Diagnosed with postural tachycardia syndrome by the Vanderbilt Autonomic - Dysfunction Center (1. increase in heart rate >/= 30 beats/minute with position change from supine to standing for 10 minutes and/or 2. Chronic symptoms consistent with POTS that are worse when upright and get better with recumbence.

Additional criteria for Control subjects:

* Healthy, non-obese, non-smokers without orthostatic tachycardia
* Selected to match profiles of POTS patients (gender, age)
* Not using vasoactive medications

Exclusion Criteria:

* Overt cause for postural tachycardia (such as acute dehydration)
* Inability to give, or withdraw informed consent
* Pregnancy
* Other factors in the investigator's opinion would prevent the subject from completing the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Postural Tachycardia Syndrome
  Controls will be age & sex matched to the patients with POTS
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
RH-PAT index | The study will be complete in approximately 2 hours. There is no follow-up to this study.
  The primary analysis of RH-PAT will involve a non-parametric, Mann Whitney U test of RH-PAT between POTS patients and Control subjects.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masuki S, Eisenach JH, Schrage WG, Johnson CP, Dietz NM, Wilkins BW, Sandroni P, Low PA, Joyner MJ. Reduced stroke volume during exercise in postural tachycardia syndrome. J Appl Physiol (1985). 2007 Oct;103(4):1128-35. doi: 10.1152/japplphysiol.00175.2007. Epub 2007 Jul 12. PMID 17626834
- [Background] Roberts LJ 2nd, Morrow JD. Isoprostanes. Novel markers of endogenous lipid peroxidation and potential mediators of oxidant injury. Ann N Y Acad Sci. 1994 Nov 15;744:237-42. doi: 10.1111/j.1749-6632.1994.tb52741.x. PMID 7825845
- [Background] Epel ES, Blackburn EH, Lin J, Dhabhar FS, Adler NE, Morrow JD, Cawthon RM. Accelerated telomere shortening in response to life stress. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17312-5. doi: 10.1073/pnas.0407162101. Epub 2004 Dec 1. PMID 15574496
- [Background] Medow MS, Minson CT, Stewart JM. Decreased microvascular nitric oxide-dependent vasodilation in postural tachycardia syndrome. Circulation. 2005 Oct 25;112(17):2611-8. doi: 10.1161/CIRCULATIONAHA.104.526764. Epub 2005 Oct 17. PMID 16230486
- [Background] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Background] Rozanski A, Qureshi E, Bauman M, Reed G, Pillar G, Diamond GA. Peripheral arterial responses to treadmill exercise among healthy subjects and atherosclerotic patients. Circulation. 2001 Apr 24;103(16):2084-9. doi: 10.1161/01.cir.103.16.2084. PMID 11319199
- [Background] Meredith IT, Currie KE, Anderson TJ, Roddy MA, Ganz P, Creager MA. Postischemic vasodilation in human forearm is dependent on endothelium-derived nitric oxide. Am J Physiol. 1996 Apr;270(4 Pt 2):H1435-40. doi: 10.1152/ajpheart.1996.270.4.H1435. PMID 8967386
- [Background] Dakak N, Husain S, Mulcahy D, Andrews NP, Panza JA, Waclawiw M, Schenke W, Quyyumi AA. Contribution of nitric oxide to reactive hyperemia: impact of endothelial dysfunction. Hypertension. 1998 Jul;32(1):9-15. doi: 10.1161/01.hyp.32.1.9. PMID 9674631
- [Background] Higashi Y, Sasaki S, Nakagawa K, Matsuura H, Kajiyama G, Oshima T. A noninvasive measurement of reactive hyperemia that can be used to assess resistance artery endothelial function in humans. Am J Cardiol. 2001 Jan 1;87(1):121-5, A9. doi: 10.1016/s0002-9149(00)01288-1. PMID 11137850
- [Background] Wilkinson IB, Qasem A, McEniery CM, Webb DJ, Avolio AP, Cockcroft JR. Nitric oxide regulates local arterial distensibility in vivo. Circulation. 2002 Jan 15;105(2):213-7. doi: 10.1161/hc0202.101970. PMID 11790703
- [Background] Noon JP, Haynes WG, Webb DJ, Shore AC. Local inhibition of nitric oxide generation in man reduces blood flow in finger pulp but not in hand dorsum skin. J Physiol. 1996 Jan 15;490 ( Pt 2)(Pt 2):501-8. doi: 10.1113/jphysiol.1996.sp021161. PMID 8821146
- [Background] Nohria A, Gerhard-Herman M, Creager MA, Hurley S, Mitra D, Ganz P. Role of nitric oxide in the regulation of digital pulse volume amplitude in humans. J Appl Physiol (1985). 2006 Aug;101(2):545-8. doi: 10.1152/japplphysiol.01285.2005. Epub 2006 Apr 13. PMID 16614356
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Dupont WD, Plummer WD. PS power and sample size program available for free on the internet. Control Clin Trials 1997;18:274
- [Derived] Chopoorian AH, Wahba A, Celedonio J, Nwazue V, Smith EC, Garland EM, Paranjape S, Okamoto LE, Black BK, Biaggioni I, Raj SR, Gamboa A. Impaired Endothelial Function in Patients With Postural Tachycardia Syndrome. Hypertension. 2021 Mar 3;77(3):1001-1009. doi: 10.1161/HYPERTENSIONAHA.120.16238. Epub 2021 Jan 25. PMID 33486983